CLINICAL TRIAL: NCT02977065
Title: Multicenter, Parallel-group, Double-blind, Randomized, Active-controlled, Dose-ranging Study to Assess the Safety, Efficacy, and Tolerability of CKD-519, Administered With HMG-CoA Reductase Inhibitors, in Subjects With Dyslipidemia
Brief Title: To Assess the Safety, Efficacy and Tolerability of CKD-519, Administered With HMG-CoA Reductase Inhibitors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 148HL16011
Record Dates: First submitted 2016-11-27; First posted 2016-11-30 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Dyslipidemias
Keywords: Dyslipidemia; CETP Inhibitors; Hyperlipidemia
MeSH Terms: conditions — Dyslipidemias; Hyperlipidemias | interventions — Atorvastatin; CKD-519; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Atorvastatin 20 mg (Active Comparator): To administrate Atorvastatin 20 mg and 4 Placebos, PO, QD for 4weeks
  Interventions: Drug: Atorvastatin 20mg
- Atorvastatin 20 mg + CKD-519 50 mg (Experimental): To administrate Atorvastatin 20 mg, CKD-519 50 mg and 3 Placebos, PO, QD for 4weeks
  Interventions: Drug: Atorvastatin 20 mg + CKD-519 50 mg
- Atorvastatin 20 mg + CKD-519 100 mg (Experimental): To administrate Atorvastatin 20 mg, CKD-519 100 mg and 3 Placebos, PO, QD for 4weeks
  Interventions: Drug: Atorvastatin 20 mg + CKD-519 100 mg
- Atorvastatin 20 mg + CKD-519 200 mg (Experimental): To administrate Atorvastatin 20 mg, CKD-519 200 mg and 2 Placebos, PO, QD for 4weeks
  Interventions: Drug: Atorvastatin 20 mg + CKD-519 200 mg
- Rosuvastatin 10 mg (Active Comparator): To administrate Rosuvastatin 10 mg and 4 Placebos, PO, QD for 4weeks
  Interventions: Drug: Rosuvastatin 10 mg
- Rosuvastatin 10 mg + CKD-519 100 mg (Experimental): To administrate Rosuvastatin 10 mg, CKD-519 100 mg and 3 Placebos, PO, QD for 4weeks
  Interventions: Drug: Rosuvastatin 10 mg + CKD-519 100 mg

INTERVENTIONS:
Drug: Atorvastatin 20mg — PO daily for 4weeks
  Other Names: Lipitor 20mg
  Arms: Atorvastatin 20 mg
Drug: Atorvastatin 20 mg + CKD-519 50 mg — PO daily for 4weeks
  Other Names: Lipitor 20mg
  Arms: Atorvastatin 20 mg + CKD-519 50 mg
Drug: Atorvastatin 20 mg + CKD-519 100 mg — PO daily for 4weeks
  Other Names: Lipitor 20mg
  Arms: Atorvastatin 20 mg + CKD-519 100 mg
Drug: Atorvastatin 20 mg + CKD-519 200 mg — PO daily for 4weeks
  Other Names: Lipitor 20mg
  Arms: Atorvastatin 20 mg + CKD-519 200 mg
Drug: Rosuvastatin 10 mg — PO daily for 4weeks
  Other Names: Crestor 10mg
  Arms: Rosuvastatin 10 mg
Drug: Rosuvastatin 10 mg + CKD-519 100 mg — PO daily for 4weeks
  Other Names: Crestor 10mg
  Arms: Rosuvastatin 10 mg + CKD-519 100 mg

SUMMARY:
A multicenter, double-blind, parallel-group, active-controlled, dose-ranging study to assess the safety and efficacy of the novel cholesteryl ester transfer protein (CETP) inhibitor CKD-519 in combination with atorvastatin or rosuvastatin in subjects with dyslipidemia.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety, efficacy, and tolerability of CKD-519, administered with HMG-CoA reductase inhibitors in subjects with dyslipidemia

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80 years.
2. Dyslipidemia with LDL-C

   * At screening if untreated: 100 to 190 mg/dL
   * At screening if treated with statins or other lipid-lowering drugs: 100 to 170 mg/dL
   * At start of double-blind treatment: 100 to 190 mg/dL.
3. HDL-C <45 mg/dL (males) or <50 mg/dL (females).
4. Fasting TG <400 mg/dL.
5. Presence of the following conditions is permitted but not mandatory, at the discretion of the investigator:

   * Treated and stable coronary heart disease without acute events in the past 3 months and stable, state-of-the-art medication.
   * Treated and stable carotid artery disease or peripheral arterial disease on stable, standard medication for the past 3 months
   * Treated and stable Type 2 diabetes mellitus with glycosylated hemoglobin (HbA1c) ≤9.5%.
6. Willing and able to sign the informed consent form (ICF).

Exclusion Criteria:

1. Chronic heart failure as defined by New York Heart Association classes III and IV.
2. Uncontrolled cardiac arrhythmias.
3. Myocardial infarction, percutaneous coronary intervention, coronary artery bypass graft, or unstable angina in past 3 months before Visit 1.
4. Stroke or transient ischemic attack within 3 months before Visit 1.
5. Uncontrolled hypertension.
6. Clinically significant laboratory abnormalities

   * Aspartate aminotransferase or alanine aminotransferase >2 times upper limit of normal range
   * Bilirubin >1.5 times upper limit of normal range
   * Creatine kinase >2 times upper limit of normal range.
7. Any active nephropathy or estimated glomerular filtration rate <60 mL/min/1.73m2 or on kidney dialysis.
8. Poorly controlled (thyroid-stimulating hormone [TSH] >2 times upper limit of normal) hyperthyroidism.
9. Homozygous familial hypercholesterolemia.
10. Intolerance or hypersensitivity to atorvastatin or rosuvastatin.
11. Prior treatment with any CETP inhibitor.
12. Positive for human immunodeficiency virus (HIV) positive, hepatitis B or hepatitis C.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline (Visit 3) in LDL-C | at Week 4

SECONDARY OUTCOMES:
Percentage change from baseline in HDL-C | at Weeks 2 and Week 4
Percentage change from baseline in concentration of HDL particles (HDL-P) | at Weeks 2 and 4
Change from baseline in size of HDL particles (HDL-P) | at Weeks 2 and 4
Percentage change from baseline in LDL-C | at Week 2
Change in concentration from baseline in LDL-C | at Weeks 2 and 4
Change in concentration from baseline in HDL-C | at Weeks 2 and 4
Percentage change from baseline in total cholesterol, TG, and non-HDL-C | at Weeks 2 and 4
Change in concentration from baseline in total cholesterol, TG, and non-HDL-C | at Weeks 2 and 4
Percentage change from baseline in apolipoprotein B (Apo B), apolipoprotein A1 (Apo A1), and apolipoprotein E (Apo E) | at Weeks 2 and 4
Change in concentration from baseline in Apo B, Apo A1, and Apo E | at Weeks 2 and 4
Percentage change from baseline in lipoprotein(a) (Lp-a) | at Weeks 2 and 4
Change in concentration from baseline in Lp-a | at Weeks 2 and 4
Change in concentration from baseline in high-sensitivity C-reactive protein at | at Weeks 2 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Mi Park, PhD, Study Director — Chong Kun Dang Pharm.
Locations (1):
- Not provided, Adelaide, Australia

IPD SHARING:
Plan to Share IPD: No